CLINICAL TRIAL: NCT00381862
Title: A Multi-Center, Trial to Evaluate the Efficacy & Tolerability of Aprepitant and Palonosetron for the Prevention of CINV in Colorectal Cancer (CRC) Patients Receiving FOLFOX
Brief Title: Phase II Trial of Aprepitant & Palonosetron for CINV Prevention w FOLFOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000503649; OHSU-SOL-06006-LM (Other: OHSU Knight Cancer Institute); OHSU-IRB-2302 (Other: OHSU IRB)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer; Nausea and Vomiting
Keywords: nausea and vomiting; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Nausea; Vomiting; Colonic Neoplasms; Rectal Neoplasms | interventions — Aprepitant; L 758298; Dexamethasone; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aprepitant and Palonosetron (Experimental)
  Interventions: Drug: aprepitant; Drug: dexamethasone; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin; Drug: palonosetron hydrochloride; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: aprepitant — Aprepitant 125 mg by mouth (PO) on day 1 and 80 mg PO on days 2 and 3 of each chemotherapy cycle
  Other Names: Emend; MK-869; L-758,298; L-754,030
Drug: dexamethasone — Dexamethasone 12 mg PO on 1st day of study drug and 8 mg PO on days 2-4
Drug: fluorouracil — as per institutional standard of care
  Other Names: 5-FU
Drug: irinotecan hydrochloride — as per institutional standard of care
  Other Names: Trade names: Camptosar®; Other names: Camptothecin-11, CPT-11
Drug: leucovorin calcium — as per institutional standard of care
  Other Names: Generic Name: Leucovorin; Other Names: Citrovorum Factor, Folinic Acid
Drug: oxaliplatin — as per institutional standard of care
  Other Names: Trade Name: Eloxatin
Drug: palonosetron hydrochloride — Palonosetron 0.25 mg IV push on day 1 only.
  Other Names: Aloxi
Procedure: quality-of-life assessment — baseline

SUMMARY:
RATIONALE: Aprepitant, palonosetron, and dexamethasone may help lessen or prevent nausea and vomiting in patients receiving chemotherapy.

PURPOSE: This phase II trial is studying how well giving aprepitant together with palonosetron and dexamethasone works in preventing nausea and vomiting caused by chemotherapy in patients receiving chemotherapy for metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy, in terms of nausea and vomiting control, of aprepitant, palonosetron hydrochloride, and dexamethasone, in preventing chemotherapy-induced nausea and vomiting in patients receiving FOLFOX or FOLFIRI chemotherapy for metastatic colorectal cancer.

Secondary

* Assess the percentage of patients with no emesis and no rescue therapy when treated with aprepitant, palonosetron hydrochloride, and dexamethasone during repeated courses of FOLFOX or FOLFIRI chemotherapy.
* Assess the effects of aprepitant on nausea, appetite, taste changes (via visual analogue scale), nutritional intake, and mucositis in these patients.
* Assess the safety of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Beginning 1 hour prior to the initiation of chemotherapy on day 1, patients receive oral aprepitant on days 1-3, oral dexamethasone on days 1-4, and palonosetron hydrochloride IV on day 1.

Nausea is assessed daily for up to 4 courses of chemotherapy.

Quality of life is assessed at baseline.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer
* Metastatic disease
* Scheduled to receive 1 of the following chemotherapy regimens*:

  * FOLFOX 4 (oxaliplatin, fluorouracil, leucovorin calcium)
  * FOLFOX 6
  * FOLFOX 7
  * FOLFIRI (irinotecan hydrochloride, fluorouracil, leucovorin calcium) NOTE: *Regimens may also include cetuximab or bevacizumab
* No emesis and no requirement for antiemetic agents within 48 hours prior to beginning chemotherapy

  * Single-agent benzodiazepines as a hypnotic allowed
* No chronic nausea

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 4 months
* White Blood Cell(WBC)count > 3,000/mm^³
* Absolute neutrophil count (ANC) > 1,500/mm^³
* Platelet count > 100,000/mm^³
* Bilirubin ≤ 2.5 times upper limit of normal (ULN) (< 5 times ULN if liver metastases present)
* Creatinine ≤ 1.5 times ULN
* Aspartate aminotransferase(AST) or Alanine aminotransferase (ALT) ≤ 2.5 times ULN (< 5 times ULN if liver metastases present)
* Able to swallow tablets and capsules
* No known sensitivity to aprepitant, palonosetron hydrochloride, or dexamethasone
* Not pregnant or nursing
* Negative pregnancy test
* No history of consuming ≥ 5 alcoholic drinks/day within the past year
* No concurrent illness requiring systemic corticosteroids other than planned dexamethasone during study treatment
* No clinical signs of active systemic infection involving the gastrointestinal tract
* No active bowel obstruction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy > Hesketh level 3

  * Prior fluorouracil with or without leucovorin calcium or capecitabine allowed
* At least 30 days since prior investigational drugs
* At least 14 days since prior neurokinin-1 antagonists
* Concurrent hydrocortisone at physiologic replacement doses (≤ 30 mg/day) allowed
* No concurrent chronic antiemetic agents
* Concurrent hypnotics allowed
* Concurrent rescue antiemetics allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, BCPS, BCOP, Study Chair — OHSU Knight Cancer Institute
Locations (6):
- United States (6):
  - St. Josephs/Cander Hospital, Savannah, Georgia
  - Kaiser Permanente, Hilo, Hawaii
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Kansas City Cancer Center, Kansas City, Missouri
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Texas A & M university / Scott and White Clinic, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant and Palonosetron: Aprepitant: 125 mg by mouth (PO) on day 1 and 80 mg PO on days 2 and 3 of each chemotherapy cycle
  Palonosetron: 0.25 mg IV push on day 1 only
Period: Overall Study
Arm/Group | Aprepitant and Palonosetron
Started | 54
Completed | 44
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Aprepitant and Palonosetron
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.728)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Emesis and no Rescue Therapy Within 5 Days of Receiving FOLFOX and FOLFIRI in the First Cycle of Chemotherapy.
Time Frame: Up to 24 weeks
Measure: Number; unit: Participants
Arm/Group | Aprepitant and Palonosetron
Number analyzed (Participants) | 54
Participants | 54

2. Secondary Outcome: Percentage of Patients With no Emesis and no Rescue Therapy During Repeated Courses of Chemotherapy
Time Frame: Duration of time that the patient is on study
Reporting Status: Not Posted

3. Secondary Outcome: Effects of Aprepitant on Nausea, Appetite, Taste Changes, (Via Visual Analogue Scale [VAS]), Nutritional Intake, and Mucositis in the Colorectal Cancer (CRC) Population.
Time Frame: Duration of time the patient is on study
Reporting Status: Not Posted

4. Secondary Outcome: To Assess the Safety of the Combination of Aprepitant, Palonosetron, and Dexamethasone in the Colorectal Cancer(CRC) Population in the First and Subsequent Cycles of Chemotherapy.
Time Frame: Duration of time patient is on study
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Patients With no Emesis and no Rescue Therapy Within 5 Days of the First Course of Chemotherapy
Time Frame: within 5 days of chemotherapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aprepitant and Palonosetron
Serious Adverse Events (participants affected / at risk) | 29/54
Other Adverse Events (participants affected / at risk) | 18/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant and Palonosetron (N=54)
Abdominal Pain (Gastrointestinal disorders) | 3 (10)
Anemia (Blood and lymphatic system disorders) | 1 (11)
Bowel Obstruction (Gastrointestinal disorders) | 1 (2)
Compression Fracture (Musculoskeletal and connective tissue disorders) | 1
Decreased Mental Status (Psychiatric disorders) | 1 (3)
Dehydration (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1 (26)
Diverticulitis (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1
GI Perforation (Gastrointestinal disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1 (7)
Hypokalemia (Blood and lymphatic system disorders) | 2 (7)
Infections (Infections and infestations) | 1 (13)
Melena (Gastrointestinal disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4 (21)
Rash (Skin and subcutaneous tissue disorders) | 2 (10)
Syncope (Vascular disorders) | 1
Transient Ischemic Attack (TIA) (Vascular disorders) | 1
Venous Thromboembolism (VTE) (Vascular disorders) | 1 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant and Palonosetron (N=54)
Fatigue (General disorders) | 7 (24)
Heartburn/ Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 3 (10)
Neuropathy-Cold Related (Nervous system disorders) | 3 (11)
Neuropathy-Peripheral/Sensory (Nervous system disorders) | 5 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No